CLINICAL TRIAL: NCT00457301
Title: An Assessment of the Effects of the Use of Measures of Health-related Quality of Life in Routine Clinical Care:an Application to Lung Transplantation.
Brief Title: Using Health-related Quality of Life (HRQL) in Routine Clinical Care
Status: Completed | Type: Observational
Sponsor: University of Alberta (Other)
Collaborators: Institute of Health Economics, Canada (Other); Roche Pharma AG (Industry)
Responsible Party: Maria Jose Santana, Lung transplant program University of Alberta Hospital
Other Study IDs: IHE-188
Record Dates: First submitted 2007-04-04; First posted 2007-04-06 (Estimated); Results first posted 2009-09-22 (Estimated); Last update posted 2020-04-01 (Actual); Status verified 2020-03

CONDITIONS: Chronic Obstructive Pulmonary Disease; Pulmonary Fibrosis; Pulmonary Hypertension; Cystic Fibrosis
Keywords: Lung transplantation, health-related quality of life.
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Pulmonary Fibrosis; Hypertension, Pulmonary; Cystic Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Control
  Interventions: Behavioral: HUI score card

INTERVENTIONS:
Behavioral: HUI score card — Patients completed the HUI2 and HUI3 before the encounter with the clinician, the result was graphically represented in the HUI score card. Clinicians used the HUI score card as an extra tool to help them in the management of the patients
  Other Names: Health Utilities Index Score Card

SUMMARY:
The objective of this study is to assess the effects of using HRQL measures in the clinical care of pre- and post-lung transplant patients.

The hypotheses are that the inclusion of HRQL measures, the Health Utilities Index System Mark 2(HUI2) and Mark 3 (HUI3), in routine clinical care of pre- and post-lung transplant patients, will: 1) improve patient-clinician communication;2) affect patient management; 3) improve patients' HRQL.

DETAILED DESCRIPTION:
Recently there has been increasing interest in the use of health-related quality of life (HRQL) measures in routine clinical practice. Traditionally, patient care has been based on laboratory results, medical history, and signs and symptoms diagnosed by clinicians. The inclusion of HRQL measures in routine practice may provide important and often otherwise missing information, revealing the impact of the disease or its treatment on the patient's physical, emotional and social well-being, and may assist in patient management. HRQL assessments may assist in changing the medical paradigm from a disease-centered approach to a patient-centered one.

Several studies in mental health and oncology discuss the application of HRQL measures in clinical practice. Taenzer et al (2000) and Detmar et al. (2002) provide evidence that using HRQL measures improves patient-clinician communication. Velikova et al (2004) detected impacts on communication and the emotional well-being of patients.

Using a framework based on these previous studies and the methods for the health technology assessment of diagnostic technologies (Guyatt et al. 1986), we will assess the effects of including HRQL assessments in the routine clinical care of patients undergoing solid organ transplantation (lung).

We expect that the routine use of HRQL measures in clinical practice will affect patient-clinician communication, patient management, and patient outcome.

Lung transplantation trades a fatal disease (end-stage pulmonary disease) for a chance at prolonged survival and improved quality of life, albeit with immunosuppression. In this context, generic preference-based measures such as HUI2 and HUI3 are preferred to specific measures, because they measure a broader range of health dimensions, including pain, ambulation and emotional issues that are expected to be relevant. Preference-based measures provide scores on the conventional 0.00 (dead) to 1.00 (perfect health) scale that allows for the integration of morbidity and mortality effects and calculation of quality adjusted life years (QALYs) and health-adjusted life expectancy (HALE).

ELIGIBILITY:
Inclusion Criteria:

* pre-lung transplant:subjects who are included on the waiting list and are being seen at the out-patient clinic
* post-lung transplant subjects.

Exclusion Criteria:

* younger than 18 years of age
* diagnosed as being cognitively impaired
* unable to complete questionnaires in English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 213 (Actual)
Dates: Start 2005-07; Primary Completion 2007-04 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David H Feeny, PhD, Principal Investigator — Professor Economics, University of Alberta
Locations (1):
- University of Alberta Hospital, Edmonton, Alberta, Canada

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment started July 2005. Patients were recruited at the out patient clinic University of Alberta Hospital.
Pre-assignment Details: Pre-transplant patients were censored out of the study once they had the lung transplant.
Groups:
- HUI2 and HUI3 Completion Without Feedback to Clinicians.: Patients in the control arm completed the HUI2 and HUI3 but the results were not fed back to clinicians.
- HUI2 and HUI3 Completion and Feedback to Clinicians: Patients in the intervention arm completed the HUI2 and HUI3 and results were fedback to clinicians before the encounter with the patient at every clinic visit.
Period: Overall Study
Arm/Group | HUI2 and HUI3 Completion Without Feedback to Clinicians. | HUI2 and HUI3 Completion and Feedback to Clinicians
Started | 105 | 108
Completed | 82 | 84
Not Completed | 23 | 24
Not completed — Withdrawal by Subject | 3 | 3
Not completed — Censored out of the study | 15 | 14
Not completed — Death | 5 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | HUI2 and HUI3 Completion Without Feedback to Clinicians. | HUI2 and HUI3 Completion and Feedback to Clinicians | Total
Number analyzed (Participants) | 105 | 108 | 213
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.4 (12.9) | 53.2 (12.6) | 53.3 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53 | 56 | 109
  Male | 52 | 52 | 104

OUTCOME MEASURES:

1. Primary Outcome: Communication Score
Description: Each clinician-patient encounter was audio tape-recorded. The content of the tape-recordings was examined and results recorded on the communication form by three blinded raters. This form tallies the number of issues discussed. The number of issues is summed to produce a communication score. The issues discussed included health attributes included in the HUI2 and HUI3: ambulation, self-care, anxiety, depression, cognitive problems, pain (type and frequency), vision, hearing speech and dexterity problems.
Time Frame: Baseline and end of study (6 months)
Population: Traditional analysis of covariance, ANCOVA was conducted to explore the difference between control and intervention groups at 6 months adjusting for baseline scores and transplant status. ITT was conducted and missing values were imputed using the LOCF.
Measure: Mean (Standard Deviation); unit: Mean number of issues discussed
Arm/Group | HUI2 and HUI3 Completion Without Feedback to Clinicians. | HUI2 and HUI3 Completion and Feedback to Clinicians
Number analyzed (Participants) | 105 | 108
Mean number of issues discussed
  baseline | 1.14 (1.16) | 1.50 (1.10)
  End-of-study | 1.36 (1.00) | 1.75 (1.15)
Statistical Analysis 1: Comparison: HUI2 and HUI3 Completion Without Feedback to Clinicians. vs HUI2 and HUI3 Completion and Feedback to Clinicians; Sample size was calculated based on the EQ-5D index score. To compare two independent means for a parallel trial design, 100 patients in each group were needed to detect a clinically important difference (CID) in EQ-5D index score (CID = 0.10, SD = 0.25) with a 5% probability of Type I error and 80% power; Test type: Superiority or Other; p = 0.05, ANCOVA; Slope = 0.28, Standard Error of Mean 0.10

2. Secondary Outcome: The Hospital Anxiety and Depression Scale,HADS. Completed at Baseline and End of the Study.
Description: HADS is a self-complete mental health measure. The scale consists of 14 items, seven of which assess anxiety and seven which assess depression. Each item is on a four point scale and the scores are added to give a total ranging from 0 to 21 for anxiety and 0 to 21 for depression. Higher scores indicate more severe anxiety or depression. A cut-point of 8 or 9 indicates mild burden for the two scales; 11 or 12 indicates severe . All the patients completed HADS at baseline and at the end of the study.
Time Frame: Baseline and end of study (6 months)
Population: 47 observation were imputed by LOCF and analyzed as ITT.
Measure: Mean (Standard Deviation); unit: mean anxiety and depression
Arm/Group | HUI2 and HUI3 Completion Without Feedback to Clinicians. | HUI2 and HUI3 Completion and Feedback to Clinicians
Number analyzed (Participants) | 105 | 108
mean anxiety and depression
  Baseline anxiety | 6.41 (3.15) | 5.81 (3.95)
  Baseline depression | 4.87 (3.48) | 4.31 (3.25)
  End-of-Study Anxiety | 5.70 (3.36) | 5.69 (3.62)
  End-of-Study Depression | 4.21 (3.71) | 4.07 (3.61)
Statistical Analysis 1: Comparison: HUI2 and HUI3 Completion Without Feedback to Clinicians. vs HUI2 and HUI3 Completion and Feedback to Clinicians; ANCOVA adjuusting for baseline HADS anxiety scores; Test type: Superiority or Other; p = 0.34, ANCOVA
Statistical Analysis 2: Comparison: HUI2 and HUI3 Completion Without Feedback to Clinicians. vs HUI2 and HUI3 Completion and Feedback to Clinicians; ANCOVA adjusting for baseline HADS depression scores; Test type: Superiority or Other; p = 0.55, ANCOVA

3. Primary Outcome: Management Composite
Description: Changes in clinical management were recorded in the chart review form. The number of referrals to other healthcare providers, tests ordered (X-rays, blood test, bronchoscopies) and changes in medication (reduction or increase dosage, addition or discontinuation) were summed to produce the management composite.
Time Frame: At baseline and end of study (6 months)
Population: Analysis was conducted using ITT, with 47 observations carried forward.
Measure: Mean (Standard Deviation); unit: mean management composite
Arm/Group | HUI2 and HUI3 Completion Without Feedback to Clinicians. | HUI2 and HUI3 Completion and Feedback to Clinicians
Number analyzed (Participants) | 105 | 108
mean management composite
  Baseline | 0.70 (1.52) | 1.20 (2.50)
  End-of-study | 2.19 (2.84) | 3.27 (3.35)
Statistical Analysis 1: Comparison: HUI2 and HUI3 Completion Without Feedback to Clinicians. vs HUI2 and HUI3 Completion and Feedback to Clinicians; Test type: Superiority or Other; p = 0.001, ANCOVA; Slope = 0.79, Standard Error of Mean 0.23

4. Primary Outcome: EuroQol, EQ-5D.
Description: Generic preference-based measure. EQ-5D consists of two sections: a 100-point visual analog scale (VAS) and a descriptive system that contains five attributes (mobility, self-care, usual activities, pain or discomfort, and anxiety or depression) with three levels per attribute ("no problem", "some problems" and "extreme problems").Using the US scoring function EQ-5D index scores range from -0.11 (all-worst health state, worse than dead), to 0.00 (dead) to 1.00 (perfect health). The EQ-5D is easy to complete, valid and reliable.
Time Frame: At baseline and end of study (6 months).
Population: To compare two independent means for a parallel trial design, 100 patients in each group were needed to detect a clinically important difference (CID) in EQ-5D index score (CID = 0.10, SD = 0.25) with a 5% probability of Type I error, two-sided-test and 80% power. ITT was conducted for 213 recruited patients. 47 records were imputed using LOCF.
Measure: Mean (Standard Deviation); unit: mean EQ-5D index score
Arm/Group | HUI2 and HUI3 Completion Without Feedback to Clinicians. | HUI2 and HUI3 Completion and Feedback to Clinicians
Number analyzed (Participants) | 105 | 108
mean EQ-5D index score
  baseline | 0.76 (0.17) | 0.76 (0.17)
  end of study | 0.75 (0.23) | 0.72 (0.25)
Statistical Analysis 1: Comparison: HUI2 and HUI3 Completion Without Feedback to Clinicians. vs HUI2 and HUI3 Completion and Feedback to Clinicians; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.46, ANCOVA; Slope = 0.01, Standard Error of Mean 0.02

ADVERSE EVENTS:
Arm/Group | HUI2 and HUI3 Completion Without Feedback to Clinicians. | HUI2 and HUI3 Completion and Feedback to Clinicians
Serious Adverse Events (participants affected / at risk) | 0/105 | 0/108
Other Adverse Events (participants affected / at risk) | 0/105 | 0/108

LIMITATIONS AND CAVEATS:
Randomizing patients instead of clinicians lead to sensitizing effects. EQ-5D is a generic preference-based measure, a specific measure should have been used to maximize responsiveness.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No